CLINICAL TRIAL: NCT05685849
Title: Valuation of Maternal Fetal Cardiac Structure and Function in Pregnancies With Cardiovascular Disease：a Prospective, Multicenter, Clinical Trial
Brief Title: Evaluation of Maternal Fetal Cardiac Structure and Function in Pregnancies With Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: MF-CAD
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy
Keywords: Pregnancy; Cardiovascular disease; Cardiac function
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial group: A total of 200 pregnant women in the first trimester (gestational age of 6-13 weeks+6 days), who had cardiovascular disease and experienced regular obstetric examinations throughout the pregnancy, were selected from the obstetric outpatients in 10 centers, with 20 cases in each center.
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — Maternal and fetal echocardiography：Time points for heart image acquisition in pregnant women: As per the Guidelines for Pre-pregnancy and Pregnancy Health Care (2018) formulated by the Obstetrics Group of the Gynecology Branch of the Chinese Medical Association, a total of five echocardiographic examinations will be performed in the first trimester(11-14 weeks of gestation), the second trimester(20-24 weeks of gestation), the third trimester(29-32 weeks of gestation), prenatal term (37-40 weeks of gestation), and 3-6 months after delivery. Time points for fetal heart image acquisition: Fetal heart images will be collected in the second trimester(20 to 24 weeks of gestation).

SUMMARY:
The First Affiliated Hospital of China Medical University initiated a multi-center study to evaluate the changes of maternal fetal heart structure and function in pregnancies with cardiovascular disease by echocardiography, to explore the impact of cardiovascular disease on maternal fetal heart, so as to provide an important reference for obstetric pregnancy risk stratification and management.

DETAILED DESCRIPTION:
Globally, the incidence rate of pregnancy with cardiovascular disease is about 1-4%, and about 15% of maternal deaths are caused by pregnancy with cardiovascular disease related complications. With the opening of China's three children policy and the increase of older mothers, the proportion of maternal deaths caused by pregnancy combined with cardiovascular disease has increased year by year, which has become the primary cause of death of critically ill pregnancies in China. In addition, maternal cardiovascular disease is also the cause of fetal growth and development, cardiac structure abnormalities, and myocardial function damage. Therefore, early sensitive detection of changes in maternal and fetal cardiac structure and function during pregnancy, accurate risk assessment of pregnancy, detailed risk stratification, timely intervention and early evaluation of therapeutic efficacy can greatly reduce maternal mortality and ensure maternal and fetal safety.

Echocardiography is the preferred method for maternal fetal heart examination during pregnancy, because it is safe and convenient, and has no radiation risk to pregnancies and fetus. It can accurately and quickly measure and evaluate cardiac cavity size, hemodynamic changes and cardiac function, and can timely detect changes in the structure and function of pregnancies and fetuses at an early stage, and conduct continuous follow-up and close monitoring in different periods of pregnancy. In recent years, most of the domestic and foreign studies on the evaluation of echocardiography in pregnancy with cardiovascular disease are single center, small sample studies, mostly for a single disease, and the follow-up time is short. Some research results are contradictory and controversial, which can not accurately reflect the maternal fetal heart changes in pregnancy with cardiovascular disease. Therefore, it is urgent to conduct a large sample, multi-center study on the evaluation of cardiovascular disease in pregnancy by echocardiography in order to provide important reference and value for the stratification and management of pregnancy risk.

In conclusion, this study used echocardiography to evaluate the changes of maternal and fetal cardiac structure and function in pregnancies with cardiovascular disease, and to explore the impact of cardiovascular disease on maternal and fetal cardiac structure and function, so as to provide an important reference for obstetric pregnancy risk stratification and management, and help clinical monitoring and management of pregnancy with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first trimester；
* 20-45 years;
* Complicated with cardiovascular diseases (mainly including congenital heart disease, aortic disease, valvular heart disease, coronary artery disease, cardiomyopathy, arrhythmia, hypertension, venous thromboembolism and other cardiovascular diseases).

Exclusion Criteria:

* Other serious diseases of the immune, respiratory, digestive, nervous, urinary, blood, endocrine and other systems;
* Tumors;
* The poor quality of ultrasound images cannot meet the requirements of parameter measurement and analysis.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: A total of 200 pregnant women in the first trimester (gestational age of 6-13 weeks+6 days), who had cardiovascular disease and experienced regular obstetric examinations throughout the pregnancy, were selected from the obstetric outpatients in 10 centers, with 20 cases in each center.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | From 11 weeks of gestation to 3-6 months postpartum
  To Evaluate of the changes of maternal cardiac systolic function in pregnancies with cardiovascular disease

SECONDARY OUTCOMES:
left ventricular global longitudinal strain | From 11 weeks of gestation to 3-6 months postpartum
  To Evaluate of the subclinical changes of maternal cardiac systolic function in pregnancies with cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, MD, Principal Investigator — First Hospital of China Medical University
Locations (10):
- China (10):
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Dalian Municipal Women and Children's Medical Center, Dalian, Liaoning
  - Women And Children's Hospital of Jinzhou, Jinzhou, Liaoning
  - Shenyang Maternity And Child Health Hospital, Shenyang, Liaoning
  - the First Hospital of China Medical Univeristy, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - ShaanXi Province People's Hospital, Xi'an, Shaanxi
  - Weifang Maternal and Child Health Hospital, Weifang, Shandong
  - Yunnan Maternal And Child Health Care Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided